CLINICAL TRIAL: NCT04711499
Title: The Effect of Fatigue on Regional Anaesthesia Task Performance Among Anaesthetists: a Rater-blinded Randomised Controlled Crossover Trial
Brief Title: Effect of Fatigue on Regional Anaesthesia Task
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: 20AN007
Record Dates: First submitted 2020-10-23; First posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2020-09

CONDITIONS: Fatigue; Anesthesia
Keywords: regional anaesthesia; patient safety; nerve blockade; ultrasound guided needling
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fatigue Group (Experimental): The trial will recruit trainee anaesthetists of ST3 grade or higher who take part in a resident night-shift rota at Nottingham University Hospitals NHS Trust. Participants will undergo baseline psychometric testing to measure baseline mood. There will be a series of questions to ascertain levels of fatigue. All participants will then be asked to perform a standardised ultrasound-guided peripheral nerve blockade task using a high fidelity bench-top phantom model. Performance in this task will be independently assessed using a previously-validated scoring tool by two raters blinded to participant group allocation.
  Interventions: Behavioral: Fatigue
- Non Fatigued group (Active Comparator): The non fatigued group will be asked to perform the same series of questions and tasks after a night at home with no work duties or commitments
  Interventions: Behavioral: Fatigue

INTERVENTIONS:
Behavioral: Fatigue — The intervention will be assessing the participant in a fatigued state compared to a non fatigued state

SUMMARY:
The adverse effects of sleep related fatigue are significant, impacting on doctors' health, wellbeing, performance and ultimately their safety and that of their patients'.

Trainees are at an increased risk of fatigue because they routinely, and are increasingly, working long hours, and exposed to excessive and high intensity workloads. With increasing numbers of patient consultations, there is a higher risk of making poorer quality clinical decisions (i.e. decision fatigue). The excessive workloads experienced by doctors can cause fatigue through the requirement for sustained attention over long periods of time, particularly when performing complex and mentally demanding tasks. Our main objective is to study the difference between the fatigued and non-fatigued state of anaesthetists and on their ability to perform an ultrasound-guided peripheral nerve blockade task. We hypothesise that fatigue will result in a clinically significant reduction in the objective structured assessment scores of anaesthetists who are performing an ultrasound-guided peripheral nerve blockade task compared to their scores when they are non-fatigued.

ELIGIBILITY:
Inclusion Criteria:

1. Anaesthetists of ST3 grade and above with previous experience of performing an ultrasound guided peripheral nerve block.

Exclusion Criteria:

1. Previous experience of gaze control training or eye-tracking software applied to medical interventions.
2. No previous experience of performing an ultrasound guided peripheral nerve block.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
composite error scoring within a regional anaesthesia performance task | 6 months
  establish a comparison of mean composite error scores (CES) between participants in group F (fatigued state) and Group A (non-fatigued state) when performing a standardised ultrasound guided regional anaesthesia task. CES can range from 0 to 100. the higher the score the more negative the performance of the candidate.

SECONDARY OUTCOMES:
Global rating score (GRS) | 6 months
  establish a comparison of mean Global rating scale (GRS) between participants in group F (fatigued state) and Group A (non-fatigued state) when performing a standardised ultrasound guided regional anaesthesia task. The GRS ranges from a score of 7 to a score of 35. The higher the score the better the performance.
Task completion time | 6 months
  Compare the mean time in seconds taken by the participants in Group F and Group A to complete the standardised UGRA task.
Reliability of the composite error score (CES) and global rating scale (GRS) | 6 months
  calculate the intra-class correlation (ICC) and Cronbach's alpha co-efficient and their associated standard error of the mean (SEM, %).
Eye tracking metrics | 6 months
  All eye tracking-derived secondary outcome measures listed below will be calculated (and summed to create a total) for each UGRA assessment using the following pre-defined areas of interest: the ultrasound machine screen ('US screen'); their hands, the needle, the US transducer or the cadaveric model ('tools'); and any other area outside the US screen or tools ('other'). This is measures on a numerical scale on the number of times there is deviation and gaze away from the screen. The lower the number the better the performance by the candidate.

CONTACTS AND LOCATIONS:
Overall Officials: David Hewson, MBBS, Principal Investigator — University Hospitals of Nottingham

IPD SHARING:
Plan to Share IPD: No